CLINICAL TRIAL: NCT02762084
Title: Double-Blind, Randomized, Vehicle-Controlled Proof of Concept Clinical Trial of Patidegib Gel 2%, 4%, and Vehicle to Decrease the Number of Surgically Eligible Basal Cell Carcinomas in Gorlin Syndrome Patients
Brief Title: Trial of Patidegib Gel 2%, 4%, and Vehicle to Decrease the Number of Surgically Eligible Basal Cell Carcinomas in Gorlin Syndrome Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PellePharm, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pelle-926-201; 2015-004274-15 (EudraCT Number)
Record Dates: First submitted 2016-04-27; First posted 2016-05-04 (Estimated); Results first posted 2019-07-15 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Basal Cell Nevus Syndrome
Keywords: Gorlin Syndrome; Basal Cell; Nevus Syndrome; BCNS; nevoid basal cell carcinoma syndrome; Basal cell carcinoma; Hedgehog; Surgically Eligible Basal Cell Carcinomas
MeSH Terms: conditions — Basal Cell Nevus Syndrome; Carcinoma, Basal Cell | interventions — IPI-926; Drug Evaluation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Patidegib gel 2% (Experimental): Patidegib gel 2%, applied topically, twice daily for 26 weeks
  Interventions: Drug: Patidegib
- Patidegib gel 4% (Experimental): Patidegib gel 4%, applied topically, twice daily for 26 weeks
  Interventions: Drug: Patidegib
- Vehicle gel (Placebo Comparator): Vehicle gel, applied topically, twice daily for 26 weeks
  Interventions: Drug: Vehicle gel

INTERVENTIONS:
Drug: Patidegib
  Other Names: Study drug
  Arms: Patidegib gel 2%; Patidegib gel 4%
Drug: Vehicle gel
  Other Names: Placebo
  Arms: Vehicle gel

SUMMARY:
Multicenter, double-blind, randomized, vehicle-controlled study that evaluates the efficacy and safety of patidegib gel 2% and 4% in comparison with vehicle in participants at least 18 years of age that meet the diagnostic criteria for basal cell nevus syndrome (BCNS). Participants will be randomized to receive patidegib gel 2%, patidegib gel 4%, or the vehicle gel for a 26-week treatment period.

DETAILED DESCRIPTION:
Participants who meet the study entry criteria will be randomized in a 1:1:1 ratio to receive patidegib gel 2%, patidegib gel 4%, vehicle gel. One or two tubes of the assigned study drug will be dispensed to the participant at the Baseline visit. Additional tubes will be dispensed at subsequent visits through Week 22. The study drug will be applied topically to the entire face as well as to treatment-targeted surgically eligible basal cell carcinomas (SEBs) at other anatomical sites twice daily for 26 weeks of treatment.

Information on reported and observed adverse events will be obtained at each visit. An abbreviated physical examination will be performed at Baseline, Week 14, and Week 26.

At Baseline and Weeks 6, 10, 14, 18, 22, and 26, all visible basal cell carcinomas (BCCs) (excluding areas below the knees) will be identified by the Investigator, circled in ink, photographed, measured, and recorded on a body diagram. Treatment-targeted SEBs (defined as the 5 SEBs on the face and/or other anatomical areas identified at Baseline as SEBs) will be treated during the 26-week treatment phase. If a participant has 5 eligible previously untreated facial SEBs (excluding tumors on nose and eyelids) these tumors will be the participant's 5 baseline treatment-targeted SEBs and non-facial baseline SEBs will not be treated with study drug. Tumors to be measured and mapped include the 5 baseline treatment-targeted tumors as well as all other facial tumors including those on the eyelids and the nose. In addition, up to 10 non-treatment-targeted non-facial tumors will also be measured and mapped.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is from 18 to 85 years of age, inclusive.
2. The participant must provide written informed consent prior to any study procedures.
3. The participant must meet diagnostic criteria for BCNS, including the first listed major criterion below plus one additional major criterion, or the first listed major criterion below plus 2 of the minor criteria outlined below:

   Major Criteria:
   * More than 2 histologically confirmed BCCs or one under the age of 20 years
   * Odontogenic keratocysts of the jaw proven by histology
   * Three or more palmar and/or plantar pits
   * Bilamellar calcification of the falx cerebri (if less than 20 years old)
   * Fused, bifid, or markedly splayed ribs
   * First degree relative with basal cell nevus syndrome
   * Patched 1 (PTCH1) gene mutation in normal tissue

   Minor Criteria:
   * Macrocephaly
   * Congenital malformations: cleft lip or palate, frontal bossing, "coarse face", moderate or severe hypertelorism
   * Skeletal abnormalities: sprengel deformity, marked pectus deformity, or marked syndactyly of the digits
   * Radiological abnormalities: bridging of the sella turcica, vertebral anomalies such as hemivertebrae, fusion or elongation of the vertebral bodies, modeling defects of the hands and feet, or flame shaped lucencies of the hands or feet
   * Ovarian fibroma
   * Medulloblastoma
4. The participant must have a history of at least 10 BCCs in toto present at Baseline and/or treated within 24 months prior to screening.
5. The participant has at Baseline a total of at least 5 previously untreated SEBs (greatest diameter 5 millimeters [mm] or greater on the face excluding the nose and periorbital skin, 9 mm or greater on non-facial areas excluding the skin below the knees), as documented clinically by the Investigator at Baseline. Untreated is define as no previous surgical or topical or intralesional drug treatment. Previous treatment with systemically administered drugs more than 6 months prior to Baseline is not considered previous treatment as long as there was no clinical evidence of resistance to oral hedgehog (HH) pathway inhibitors (such as vismodegib, patidegib, and sonidegib). Baseline treatment-targeted SEBs must not exceed a diameter of >2 centimeters (cm). At least one of these tumors must be appropriate for a 2 mm punch biopsy for biomarker analysis at Baseline and Week 6 visits. If a participant has 5 or more facial, excluding periorbital and nasal skin, SEBs at Baseline, non-facial SEBs will not be treatment-targeted SEBs.
6. The participant is willing to have SEBs biopsied for biomarkers and plasma to be collected to measure drug levels as required in the protocol.
7. The participant is willing to abstain from application of non-study topical prescription and over the counter medications to facial skin and within 5 cm of treatment targeted SEBs at other anatomical areas for the duration of the study except as prescribed by the Investigator. Moisturizers and emollients are allowable. Participants will be encouraged to use sunscreen with a sunscreen protection factor (SPF) 15 or higher at least once daily on all exposed skin sites.
8. Female participants must have a negative serum pregnancy test at Screening.
9. If the participant is a male with a female sexual partner who is of childbearing potential the couple is willing to use two effective methods of birth control during the duration of the trial and for one month after the last application of the gel. A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (that is, has had menses at any time in the preceding 24 consecutive months), must agree to use 2 effective methods of contraception for the duration of the study and at least 1 month after the last study drug application. The two forms of birth control authorized are defined as the use of a barrier method of contraception (condom with spermicide) in association with one of the following methods of birth control: bilateral tubal ligation; combined oral contraceptives (estrogens and progesterone) or implanted or injectable contraceptives with a stable dose for at least 1 month prior to Baseline; hormonal intra-uterine device (IUD) inserted at least 1 month prior to Baseline.
10. The participant is willing to contact the study center after each primary skin care physician (PSCP) visit to provide the study center details of the visit and any treatment of skin tumors.
11. The participant is willing to forego treatment of the treatment targeted baseline SEBs except when the Investigator and/or primary care giver believes that delay in treatment potentially might compromise the health of the participant.

Exclusion Criteria:

1. The participant is a woman of childbearing potential. This proscription is based on the key role of the HH pathway in embryogenesis, the known preclinical teratogenic effects of systemic cyclopamine, a naturally occurring inhibitor of SMO, and the unknown level of systemic exposure following topical application in humans. A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (that is, has had menses at any time in the preceding 24 consecutive months).
2. The participant has used topical products to the face or within 5 cm of a treatment targeted SEB or systemic therapies that might interfere with the evaluation of the study medication during the study. Specifically, these include the use of:

   * Topical glucocorticoids 30 days prior to screening
   * Retinoids (such as etretinate, isotretinoin, tazarotene, tretinoin, adapalene) systemically or topically or > 5% of an alphahydroxy acid (such as glycolic acid, lactic acid) or 5-fluorouracil or imiquimod (except as topical treatment to discrete BCCs) systemically or topically to the skin during the 6 months prior to entry.
   * Systemic chemotherapy within one year prior to screening. (Note: field therapy with topically applied treatments can be done as long as they are not applied within 5 cm of a treatment targeted tumor).
   * Known inhibitors of the HH signaling pathway (such as vismodegib, patidegib, and sonidegib) topically or systemically within 6 months of entry into the study.
3. The participant has a history of hypersensitivity to any of the ingredients in the study drug formulation.
4. The participant is unable or unwilling to make a good faith effort to return for all follow-up visits and tests.
5. The participant has uncontrolled systemic disease.
6. The participant has clinically important history of liver disease, including viral hepatitis, current alcohol abuse, or cirrhosis.
7. The participant has any condition or situation which in the Investigator's opinion may put the participant at significant risk, could confound the study results, or could interfere significantly with the participant's participation in the study. This includes history of other skin conditions or diseases, metabolic dysfunction, physical examination findings, or clinical laboratory findings giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or render the participant at high risk from treatment complications.
8. The participant has a history of invasive cancer within the past 5 years excluding non-melanoma skin cancer, Stage I cervical cancer, ductal carcinoma in situ of breast, or chronic lymphocytic lymphoma (Stage 0).
9. The participant has current, recent (within 4 weeks of Baseline visit), or planned participation in an experimental drug study while enrolled in this study.
10. Female sexual partner(s) of male participants who are unwilling or unable to comply with pregnancy prevention measures.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2017-04-24 (Actual); Study Completion 2017-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Lear, MD, Principal Investigator — Manchester Royal Infirmary
Locations (2):
- United Kingdom (2):
  - Royal London Hospital, London
  - Manchester Royal Infirmary, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Patidegib Gel 2%; Patidegib Gel 4%; Vehicle Gel: Applied topically twice daily for 26 weeks
Period: Overall Study
Arm/Group | Patidegib Gel 2% | Patidegib Gel 4% | Vehicle Gel
Started | 6 | 6 | 5
Received at Least 1 Dose of Study Drug | 6 | 6 | 5
By Tumor Per Protocol Population (PP) (All treatment-targeted tumors except those biopsied and those that did not meet protocol criteria.) | 6 | 6 | 4
Completed | 5 | 6 | 4
Not Completed | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Patidegib Gel 2% | Patidegib Gel 4% | Vehicle Gel | Total
Number analyzed (Participants) | 6 | 6 | 5 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (12.14) | 62.5 (13.87) | 58.8 (17.58) | 60.8 (13.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 3 | 11
  Male | 1 | 3 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 5 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 6 | 5 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 6 | 5 | 17
Weight [Mean (Standard Deviation); unit: kilograms] — Population: Weight data at baseline was not available for 1 participant in the Patidegib Gel 4% treatment arm.
  kilograms
    number analyzed (Participants) | 6 | 5 | 5 | 16
    (all) | 90.73 (20.539) | 81.60 (11.872) | 81.52 (21.477) | 85.00 (17.95)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Efficacy: Percent Change in Tumor Size of Treatment-targeted Surgically Eligible Basal Cell Carcinomas (SEBs) From Baseline
Description: SEBs were defined as clinically diagnosed basal cell carcinoma (BCC) 5 millimeters (mm) or greater in diameter on the face, excluding the nose and periorbital skin, and 9 mm or greater at sites other than the face. The percent change in greatest diameters of treatment-targeted surgically eligible basal cell carcinomas (SEBs) from Baseline to Week 26 was calculated as follows: (sum [Baseline] - sum [Week 26] / sum [Baseline] * 100), where sum = the greatest diameters of Baseline treatment-targeted SEBs and positive numbers represent decrease in tumor size and negative numbers to represent increase in tumor size. Missing values were imputed using Last-Observation Carried Forward (LOCF).
Time Frame: Baseline, Week 26
Population: By tumor per protocol population includes all treatment-targeted tumors except tumors that were biopsied and excludes tumors that did not meet protocol criteria.
Measure: Mean (Standard Deviation); unit: percentage change
Units Other Than Participants: Number of tumors
Arm/Group | Patidegib Gel 2% | Patidegib Gel 4% | Vehicle Gel
Number analyzed (Participants) | 6 | 6 | 4
Number analyzed (Number of tumors) | 21 | 24 | 16
percentage change | 51.29 (41.780) | 26.63 (41.270) | 21.82 (25.213)
Statistical Analysis 1: Comparison: Patidegib Gel 2% vs Vehicle Gel; at Week 26; Test type: Other — Pairwise comparison; p = 0.030, ANCOVA; ANCOVA with treatment group as a factor and Baseline value as a covariate
Statistical Analysis 2: Comparison: Patidegib Gel 4% vs Vehicle Gel; at Week 26; Test type: Other — Pairwise comparison; p = 0.756, ANCOVA; ANCOVA with treatment group as a factor and Baseline value as a covariate

2. Primary Outcome: Molecular Efficacy: Percent Change in the Hedgehog (HH) Signaling Pathway Target Gene Glioma-associated Oncogene Homolog 1 (GLI1) Messenger Ribonucleic Acid (mRNA) Levels From Baseline
Description: SEBs were defined as clinically diagnosed BCC 5 mm or greater in diameter on the face, excluding the nose and periorbital skin, and 9-mm or greater at sites other than the face. A single baseline SEB designated as a treatment targeted tumor at Baseline was biopsied first at Baseline and again following 6 weeks of treatment. This was used to assess percent change in GLI1 mRNA levels as follows: (Baseline - Week 6) / Baseline * 100, where positive numbers to represent decrease in GL1 mRNA level and negative numbers to represent increase in GL1 mRNA level. Any missing values were not imputed; all available data is summarized.
Time Frame: Baseline, Week 6
Population: Participants who received at least 1 dose of study drug who had evaluable GLI1 mRNA data at Baseline and Week 6.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Patidegib Gel 2% | Patidegib Gel 4% | Vehicle Gel
Number analyzed (Participants) | 4 | 4 | 4
percentage change | 53.83 (27.197) | 20.69 (34.730) | 28.53 (43.096)
Statistical Analysis 1: Comparison: Patidegib Gel 2% vs Vehicle Gel; at Week 6; Test type: Other — Pairwise comparison; p = 0.500, ANCOVA; ANCOVA with treatment group as a factor and using Baseline value as a covariate
Statistical Analysis 2: Comparison: Patidegib Gel 4% vs Vehicle Gel; at Week 6; Test type: Other — Pairwise comparison; p = 0.681, ANCOVA; ANCOVA with treatment group as a factor and using Baseline value as a covariate

3. Primary Outcome: Safety and Tolerability Assessment of Treatment With Patidegib Gel: Number of Participants With a Treatment-emergent Adverse Event Causally Related to Study Drug
Description: All serious adverse events (SAEs) and all other non-serious adverse events (AEs) regardless of causality are located in the Reported AE Module. AEs considered as related where categorized by the Investigator as either definitely related, probably related, or possibly related. Treatment-emergent AEs are those with an onset after use of study drug.
Time Frame: Baseline through Week 26
Population: All enrolled participants who were randomized, received at least 1 confirmed dose of study drug, and had at least 1 post-baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Patidegib Gel 2% | Patidegib Gel 4% | Vehicle Gel
Number analyzed (Participants) | 6 | 6 | 5
Participants | 2 | 5 | 2

4. Primary Outcome: Safety and Tolerability Assessment of Treatment With Patidegib Gel: Number of Participants With Treatment-emergent Administrative Site Skin Condition AEs Causally Related to Study Drug
Description: All SAEs and all other non-serious AEs, regardless of causality, are located in the Reported AE Module. The number of participants reporting administrative-site, skin condition treatment-emergent AEs considered related to study drug by the Investigator are presented below. Treatment-emergent AEs are those with an onset after use of study drug.
Time Frame: Baseline through Week 26
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Patidegib Gel 2% | Patidegib Gel 4% | Vehicle Gel
Number analyzed (Participants) | 6 | 6 | 5
participants
  Application site alopecia | 0 | 1 | 0
  Application site dermatitis | 0 | 1 | 0
  Application site pain | 0 | 1 | 0
  Application site rash | 0 | 1 | 0
  Application site reaction | 0 | 0 | 1

5. Secondary Outcome: The Number of Participants Reporting New SEBs on the Face From Baseline for the Combined Patidegib Treatment Groups
Description: Facial SEBs were defined as clinically diagnosed BCC 5 mm or greater in diameter on the face, excluding the nose and periorbital skin. A new facial SEB was defined as an SEB first noted on the face after Week 2 that developed at a site where there was no visible BCC of any size at Baseline or Week 2. New facial SEBs were investigated for participants on vehicle gel versus participants on patidegib 2% and 4% gel. Missing values were imputed using LOCF.
Time Frame: Baseline, Week 26
Population: Participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Groups:
- Patidegib Gel: Patidegib: 2% or 4% gel applied topically twice daily for 26 weeks
Arm/Group | Patidegib Gel | Vehicle Gel
Number analyzed (Participants) | 12 | 5
participants | 2 | 3

6. Secondary Outcome: The Mean Number of New SEBs on the Face for the Combined Patidegib Treatment Groups
Description: Facial SEBs were defined as clinically diagnosed BCC 5 mm or greater in diameter on the face, excluding the nose and periorbital skin. A new facial SEB was defined as an SEB first noted on the face after Week 2 that developed at a site where there was no visible BCC of any size at Baseline or Week 2. New facial SEBs were investigated for participants on vehicle gel versus participants on patidegib 2% and 4% gel. Missing values were imputed using LOCF. The mean number of new SEBs (number per participant) are presented. No measure of dispersion/precision was calculated.
Time Frame: Baseline, Week 26
Population: Participants who received at least 1 dose of study drug.
Measure: Number; unit: new SEBs
Arm/Group | Patidegib Gel | Vehicle Gel
Number analyzed (Participants) | 12 | 5
new SEBs | 0.4 | 1.4
Statistical Analysis 1: Comparison: Patidegib Gel vs Vehicle Gel; at Week 26; Test type: Other — One-sided comparison; p = 0.048, Mann Whitey U
Statistical Analysis 2: Comparison: Patidegib Gel vs Vehicle Gel; at Week 26; Test type: Other — Two-sided comparison; p = 0.096, Mann Whitey U

7. Secondary Outcome: The Mean Number of New SEBs on the Face for the Combined Patidegib Treatment Groups by Tumor Population
Description: as for outcome 6
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Number; unit: new SEBs
Arm/Group | Patidegib Gel | Vehicle Gel
Number analyzed (Participants) | 12 | 5
new SEBs | 0.3 | 1.4
Statistical Analysis 1: Comparison: Patidegib Gel vs Vehicle Gel; at Week 26; Test type: Other — Two-sided comparison; p = 0.008, Mann Whitey U

8. Secondary Outcome: Percent Change in Baseline Treatment-targeted SEBs Tumor Size From Baseline
Description: SEBs were defined as clinically diagnosed BCC 5 mm or greater in diameter on the face, excluding the nose and periorbital skin, and 9 mm or greater at sites other than the face. The percent change in greatest diameters of Baseline treatment-targeted SEBs from Baseline to Week x (Week 6, 10, 14, 18, or 22) was calculated as follows: (sum [Baseline] - sum [Week x] / sum [Baseline] * 100), where sum = the greatest diameters of Baseline treatment-targeted SEBs, and positive numbers to represent decrease in tumor size and negative numbers to represent increase in tumor size. Missing values were imputed using LOCF.
Time Frame: Baseline and Weeks 6, 10, 14, 18, and 22
Population: Participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Patidegib Gel 2% | Patidegib Gel 4% | Vehicle Gel
Number analyzed (Participants) | 6 | 6 | 5
percentage change
  Week 6 | 16.0 (37.07) | 6.1 (10.41) | 8.2 (4.55)
  Week 10 | 30.8 (39.54) | 10.7 (12.00) | 10.5 (5.35)
  Week 14 | 36.1 (46.45) | 14.1 (13.18) | 10.7 (6.26)
  Week 18 | 26.0 (73.79) | 18.4 (26.86) | 19.6 (21.98)
  Week 22 | 32.1 (78.71) | 23.2 (22.87) | 23.2 (28.03)

9. Secondary Outcome: Percent Change in Central Facial SEBs From Baseline
Description: Central facial SEBs were defined as those located on the nose or periorbital area (eyelids) which were 3 mm or greater at Baseline. The percent change from Baseline to Week x (Week x = Weeks 6, 10, 14, 18, 22, or 26) in central facial SEBs was calculated as follows: [sum (Baseline) - sum (Week x)] / [sum (Baseline)] * 100 where sum = the greatest diameters of Baseline treatment-targeted SEBs where positive numbers to represent decrease in tumor size and negative numbers to represent increase in tumor size. Missing values were imputed using LOCF.
Time Frame: Baseline and Weeks 6, 10, 14, 18, 22, and 26
Population: Participants who received at least 1 dose of study drug and who had a central facial SEB at Baseline.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Patidegib Gel 2% | Patidegib Gel 4% | Vehicle Gel
Number analyzed (Participants) | 1 | 2 | 2
percent change
  Week 6 | 5.9 (NA) — Standard deviation was not calculated because there was only 1 participant in the analysis population. | -20.0 (28.28) | 8.0 (24.11)
  Week 10 | 5.9 (NA) — Standard deviation was not calculated because there was only 1 participant in the analysis population. | -10.0 (42.43) | 12.5 (17.68)
  Week 14 | 5.9 (NA) — Standard deviation was not calculated because there was only 1 participant in the analysis population. | -60.0 (84.85) | 29.5 (28.93)
  Week 18 | 5.9 (NA) — Standard deviation was not calculated because there was only 1 participant in the analysis population. | -70.0 (70.71) | 17.0 (11.25)
  Week 22 | 5.9 (NA) — Standard deviation was not calculated because there was only 1 participant in the analysis population. | -45.0 (63.64) | 29.5 (28.93)
  Week 26 | 5.9 (NA) — Standard deviation was not calculated because there was only 1 participant in the analysis population. | -65.0 (63.64) | 20.5 (41.78)

10. Secondary Outcome: Proportion of Non-central Facial BCCs Increasing to ≥ 5 mm From Baseline
Description: The proportion of non-central facial BCCs that at Baseline measured a greatest diameter of < 5 mm and increased to a diameter of ≥ 5 mm by Week x (Week x = Weeks 6, 10, 14, 18, 22, or 26) were calculated for each participant as follows: (Number of non-central facial BCCs with greatest diameter ≥ 5 mm at Week x) / (Number of non-central facial BCCs with greatest diameter < 5 mm at Baseline). Missing values were imputed using LOCF.
Time Frame: Baseline and Weeks 6, 10, 14, 18, 22, and 26
Population: Participants who received at least 1 dose of study drug with non-central facial BCCs < 5 mm at Baseline.
Measure: Mean (Standard Deviation); unit: proportion of BCCs
Arm/Group | Patidegib Gel 2% | Patidegib Gel 4% | Vehicle Gel
Number analyzed (Participants) | 3 | 2 | 3
proportion of BCCs
  Week 6 | 0.17 (0.289) | 0 (0) | 0.17 (0.289)
  Week 10 | 0 (0) | 0.67 (0.474) | 0.17 (0.289)
  Week 14 | 0 (0) | 0 (0) | 0 (0)
  Week 18 | 0 (0) | 0.17 (0.233) | 0 (0)
  Week 22 | 0 (0) | 0.34 (0.474) | 0 (0)
  Week 26 | 0 (0) | 0 (0) | 0.11 (0.191)

11. Secondary Outcome: Proportion of Treatment-Targeted SEBs No Longer Classified as SEBs After 26 Weeks
Description: SEBs were defined as clinically diagnosed BCC 5 mm or greater in diameter on the face, excluding the nose and periorbital skin, and 9 mm or greater at sites other than the face. The proportion of Baseline treatment-targeted SEBs that at the end of 26 weeks of treatment were no longer large enough to be classified as SEBs (that is, the proportion of Baseline treatment targeted SEBs on the face that became < 5 mm in greatest diameter and non-facial Baseline treatment targeted SEBs that became < 9 mm in greatest diameter) were calculated for each participant as follows:
  (Number of Baseline treatment-targeted facial SEBs with greatest diameter < 5 mm) + (Baseline treatment targeted non-facial SEBs with greatest diameter < 9 mm) / Number of baseline treatment targeted SEBs.
  Missing values were imputed using LOCF.
Time Frame: Baseline and Weeks 6, 10, 14, 18, 22, and 26
Population: Participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: proportion of SEBs
Arm/Group | Patidegib Gel 2% | Patidegib Gel 4% | Vehicle Gel
Number analyzed (Participants) | 6 | 6 | 5
proportion of SEBs
  Week 6 | 0.37 (0.497) | 0.13 (0.242) | 0.12 (0.179)
  Week 10 | 0.40 (0.473) | 0.13 (0.103) | 0.16 (0.219)
  Week 14 | 0.53 (0.468) | 0.23 (0.234) | 0.16 (0.219)
  Week 18 | 0.57 (0.497) | 0.23 (0.320) | 0.28 (0.303)
  Week 22 | 0.53 (0.516) | 0.30 (0.276) | 0.32 (0.363)
  Week 26 | 0.53 (0.516) | 0.30 (0.303) | 0.36 (0.434)

12. Other Pre Specified Outcome: Percentage of Treatment-targeted SEBs Achieving Clear or Almost Clear on the 5-point Investigator Static Global Tumor Assessment (ISGTA) Scale
Description: The ISGTA is a scale with scores ranging from 0 (clear), 1 (almost clear), 2 (minimal residual tumor), to 3 (clearly visible tumor). The Investigator assessed each Baseline treatment-targeted SEB at Weeks 6, 10, 14, 18, 22, and 26. SEBs were defined as clinically diagnosed BCC 5 mm or greater in diameter on the face, excluding the nose and periorbital skin, and 9 mm or greater at sites other than the face. The percentage of Baseline treatment-targeted SEBs evaluated as being clear or almost clear at Week x (Week x = Week 6, 10, 14, 18, 22 or 26) based on the ISGTA scale was calculated as follows: (Number of baseline treatment-targeted SEBs with ISGTA score of 0 or 1 at Week x) / (Number of Baseline treatment-targeted SEBs) * 100. Missing data were imputed using LOCF. The percentage of responders achieving clear (0) or almost clear (1) on the ISGTA scale are presented by Week.
Time Frame: Baseline and Weeks 6, 10, 14, 18, 22, and 26
Population: Participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of SEBs
Arm/Group | Patidegib Gel 2% | Patidegib Gel 4% | Vehicle Gel
Number analyzed (Participants) | 6 | 6 | 5
percentage of SEBs
  Week 6 | 23.3 | 3.3 | 12.0
  Week 10 | 23.3 | 13.3 | 8.0
  Week 14 | 33.3 | 13.3 | 8.0
  Week 18 | 33.3 | 23.3 | 20.0
  Week 22 | 36.7 | 26.7 | 20.0
  Week 26 | 33.3 | 30.0 | 24.0

ADVERSE EVENTS:
Time Frame: 26 Weeks
Arm/Group | Patidegib Gel 2% | Patidegib Gel 4% | Vehicle Gel
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 2/5
Other Adverse Events (participants affected / at risk) | 4/6 | 6/6 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patidegib Gel 2% (N=6) | Patidegib Gel 4% (N=6) | Vehicle Gel (N=5)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patidegib Gel 2% (N=6) | Patidegib Gel 4% (N=6) | Vehicle Gel (N=5)
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Episcleritis (Eye disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0
Food Poisoning (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Application site alopecia (General disorders) | 0 | 1 | 0
Application site dermatitis (General disorders) | 0 | 1 | 0
Application site pain (General disorders) | 0 | 1 | 0
Application site rash (General disorders) | 0 | 1 | 0
Application site reaction (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 2 | 3 | 2
Candida infection (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercholesterolaemina (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Ageusia (Nervous system disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 1
Trigeminal neuralgia (Nervous system disorders) | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-05-12): https://cdn.clinicaltrials.gov/large-docs/84/NCT02762084/SAP_000.pdf
  • Study Protocol (2016-08-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT02762084/Prot_001.pdf